CLINICAL TRIAL: NCT05764174
Title: Digital Applications to Monitor Novel Coronavirus Disease and Response in Colombia - Syndromic and Vaccination Surveillance
Acronym: DIAMOND-R
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Pontificia Universidad Javeriana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 00017868
Record Dates: First submitted 2023-01-12; First posted 2023-03-10 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Vaccination Refusal; COVID-19
MeSH Terms: conditions — Vaccination Refusal; COVID-19

STUDY DESIGN:
Intervention Model Description: Three treatment arms and one control will be deployed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Factual messages (Active Comparator): Participants in the arm with factual messages will listen to actual data on vaccination.
  Interventions: Behavioral: Factual messages
- Narrative message (Active Comparator): Participants the narrative messages will listen to messages appealing to emotions that were explored in a qualitative study conducted earlier.
  Interventions: Behavioral: Narrative message
- Mixed messages (Active Comparator): The mixed arm will combine both factual and narrative messages.
  Interventions: Behavioral: Mixed message
- Control arm (No Intervention): Participants in the control arm will not be provided with a message and will only be asked for whether they participant got vaccinated in the last two weeks.

INTERVENTIONS:
Behavioral: Factual messages — Messages with descriptive data on COVID-19 vaccines
  Arms: Factual messages
Behavioral: Narrative message — Messages with emotional descriptions on COVID-19 vaccines
  Arms: Narrative message
Behavioral: Mixed message — Messages with both descriptive data and emotional descriptions on COVID-19 vaccines
  Arms: Mixed messages

SUMMARY:
Brief Summary: The main objective of this activity is to assess the effectiveness of different messaging strategies (factual, narrative, mixed and a control) to promote COVID-19 adult vaccination.

DETAILED DESCRIPTION:
The investigators deploy mobile phone surveys using Interactive Voice Response (IVR) in a random sample of mobile phone numbers (random digit dialing or RDD) in Colombia.

Adult individuals who have not been fully vaccinated against COVID-19 (defined as those who 1) did not get any vaccine; 2) did not get the complete vaccination scheme 3) did not get one booster when less than 50 years old; 4) did not get two boosters when older than 50 years old), and who consent to be recontacted are invited to participate in the messaging trial. After consent, participants are randomized in three different treatment arms or one control arm. Participants in each treatment arm are presented with different messages to improve COVID-19 vaccination. Participants in the arm with factual messages listen to actual data and scientifical information on COVID-19 vaccination. Those in the narrative arm listen to messages appealing to emotions drawing on the COVID-19 vaccination experiences that were explored in a qualitative study conducted earlier. The mixed arm combines both factual and narrative messages. Finally, the control arm does not deliver any message and will only ask for whether the participant got vaccinated in the last two weeks. Individuals in each of the three treatment arms receive seven different types of messages. Each message is delivered twice every week for seven weeks and their vaccination status is inquired in the same calls to assess whether the participants received their vaccine after the last call. IN all arms, respondents are asked a simple question to test the attention they pay to the information provided in the message. The three treatment arms are compared against the control to assess the probability that any of the arms is significantly better than the control. With this aim, the minimum target sample size for each messaging group is N=173 which allows for the detection of a difference between groups of at least 15% with a double-tailed distribution at alpha=0.05 and power =0.8.

The investigators launched a first cohort on September 21, 2022 over sampling both the treatment and control arms to reduce the risk of attrition and aiming at obtaining 250 recruited participants that agree to participate. Due to high attrition, a second cohort was deployed on October 25, 2022 following the same procedure as for the first cohort, this time with a target of 400 recruited respondents with the aim of achieving the required sample size.

The investigators assess the differential likelihood of vaccinating during the trial for individuals participating in the different arms, including the control.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the trial
* Being older than 18
* Have not been fully vaccinated against COVID-19 (those who did not get any vaccine, did not get the complete vaccination scheme or did not get one booster if less than 50 or two boosters if older than 50).

Exclusion Criteria:

* Willingness to stop their participation in the trial
* Being younger than 18
* Have been fully vaccinated against COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2409 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2022-12-17 (Actual); Study Completion 2022-12-17 (Actual)

PRIMARY OUTCOMES:
Percentage point change on the probability of new vaccination for treatment arms vs. control | 7 weeks
  The participant reports to have been vaccinated against COVID-19 in the last two weeks

SECONDARY OUTCOMES:
Percentage point change on the probability of new vaccination conditional on correct answer to the test | 7 weeks
  The participant reports to have been vaccinated against COVID-19 in the last two weeks and also has a high score on the response to the tests after the message
Percentage point change on the probability of new vaccination conditional on demographic, socioeconomic and health characteristics | 7 weeks
  The participant reports to have been vaccinated against COVID-19 in the last two weeks and that likelihood is related to specific demographic, health and socioeconomic variables captured
Percentage of attrition between each of the different waves of messages. | 7 weeks
  Participants enrolling in the trial, decide to stop participating at any time. The likelihood of participation is assessed in correlation with sociodemographic variables.

CONTACTS AND LOCATIONS:
Overall Officials: Andres Vecino, MD PhD, Principal Investigator — Johns Hopkins Bloomberg School of Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
IPD will only be analyzed by the Johns Hopkins team in an anonymized manner. Other researchers will have access only to aggregated information. No attempts to obtain identifiable information will be done and the numbers will be deleted from the main database once completed the data collection